CLINICAL TRIAL: NCT01332695
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over, Safety, Tolerability and Proof of Concept Study of ST101 for Essential Tremor
Brief Title: A Pilot Efficacy and Safety Study of ST101 in Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sonexa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST101-A002-203
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Essential Tremor
Keywords: tremor; WHIGET; Fahn Tolosa Marin Scale
MeSH Terms: conditions — Essential Tremor; Tremor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ST101 (Experimental): ST101 oval tablets
  Interventions: Drug: ST101
- Placebo (Placebo Comparator): oval tablets to match ST101 tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ST101 — tablets for oral administration
  Arms: ST101
Drug: Placebo — placebo to match
  Arms: Placebo

SUMMARY:
This study will look at the ability of ST101 to treat symptoms in subjects with Essential Tremor. This study will also examine the safety and tolerability of the drug. This study is evaluating one dose level of ST101 versus placebo in a cross-over fashion. This means that all patients will receive both ST101 and placebo, but they will receive it in a random (by chance) order.

DETAILED DESCRIPTION:
Essential tremor (ET) is a slowly progressive, chronic neurological disorder characterized by a 4- to 12-Hertz tremor, which can involve the arms, head, voice and lower extremities. Although the hallmark of the disorder is thought to be the kinetic tremor, ET patients usually also manifest a postural tremor as well. Kinetic tremor (tremor with voluntary movements) may interfere with fine motor skills (e.g., writing, eating, drinking from a cup, pouring liquids); and depending upon its severity, may result in significant disability and diminished quality of daily living. Essential tremor represents an area of unmet medical need and this study is designed as a safety, tolerability and proof-of-concept investigation of the ability of ST101 to improve tremor. In this 2-stage study, subjects will be randomly assigned to either ST101 or placebo in Stage 1, and will receive the alternate treatment in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or probable essential tremor (ET) as defined by the Tremor Investigational Group with involvement of the hands and arms of at least 2 years duration
* Tremor severity score of >/= 2 in at least one upper extremity on the Fahn-Tolosa-Marin Tremor Rating Scale
* Subject who is accessible by telephone
* Subject who can comply with study visits, study drug compliance, and study procedures.

Exclusion Criteria:

* Subject whose tremor is adequately controlled on a current treatment
* Subject who is pregnant, plans to become pregnant during the study or within 2 months of completing the study or who is presently lactating or breast-feeding
* Subject with other medical conditions that may cause or explain subject's tremor
* Subject with a recent history of hematologic/oncologic disorders
* Subject taking medication(s) that might produce tremor or interfere with the evaluation of tremor
* Subject who has had surgical intervention for their tremor in the past (e.g., ablative thalamotomy or gamma knife thalamotomy), or has had a botulinum toxin injection in the 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Washington Heights-Inwood Genetic Study of Essential Tremor (WHIGET) Rating Scale | Baseline, Week 3, Week 5, Week 8
  The WHIGET Rating Scale is a 6-item scale. Ratings are performed for the right and left side for each activity. Each subject is videotaped in the same manner performing set activities, which are then rated. Rated tasks involve fine motor skills. Each item is scored by an independent, central, blinded reader, and the item scores are summed to provide a total score. Total score range is from 0 to 48, with an increase in score reflecting an increase in ET severity.

SECONDARY OUTCOMES:
Functional Disabilities Scale | Screening, Baseline, Weeks 3, 5, 8
  An 8-Item functional scale that assesses the following functional domains: Speaking/Phonation, Feeding (other than liquids), Bringing Liquids to Mouth, Hygiene, Dressing, Writing, Working, and Social Activities. Higher scores indicate worsening of disease.
Clinical Global Impression of Change | Week 3, Week 8
  A 7-point Likert scale with Marked Worsening to Marked Improvement at the extremes, and Unchanged in the center. Scores range from -3 to +3 wherein negative scores indicate worsening, while positive scores indicate improvement.
Subject Clinical Global Impression of Change | Week 3, Week 8
  A global visual analog scale (VAS) which is a 100 mm horizontal line on which the subject indicates their overall assessment of response to study drug by making a mark on the horizontal line.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles, California, United States